CLINICAL TRIAL: NCT01190189
Title: Safety Study of GSK Biologicals' Human Papillomavirus Vaccine (GSK-580299) in Healthy Female Control Subjects From the Primary NCT00294047 Study
Brief Title: Safety Evaluation of the GSK-580299 Vaccine in Women From the Control Group in the Primary NCT00294047 Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 113621
Record Dates: First submitted 2010-08-26; First posted 2010-08-27 (Estimated); Results first posted 2018-12-17 (Actual); Last update posted 2019-06-19 (Actual); Status verified 2019-06

CONDITIONS: Infections, Papillomavirus
Keywords: Serious adverse events (SAEs); HPV vaccine; Medically significant conditions; Cervical neoplasia
MeSH Terms: conditions — Papillomavirus Infections | interventions — human papillomavirus vaccine, L1 type 16, 18

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cervarix Group (Experimental): Healthy female subjects who received control vaccine in the primary study HPV-015 (NCT00294047), were administered three doses of Cervarix vaccine intramuscularly, according to a 0,1,6-month schedule.
  Interventions: Biological: GSK580299 (Cervarix)

INTERVENTIONS:
Biological: GSK580299 (Cervarix) — 3-dose schedule intramuscularly vaccination

SUMMARY:
This extension study is designed to assess the safety of GSK Biological's human papillomavirus (HPV) vaccine GSK580299 in female subjects who took part in the primary study NCT00294047 and received the control vaccine in countries for which the licensed GSK HPV vaccine is not indicated for the subject's age group (26 years and older). This study is thus conducted to enable all women who received the control placebo in the primary NCT00294047 study to receive the GSK580299 vaccine.

DETAILED DESCRIPTION:
This Protocol Posting has been updated following Protocol Amendment 1, December 2010, leading to the update of 1 of the primary outcome measures and following Protocol Amendment 2, January 2011, leading to the removal of one of the exclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes can and will comply with the requirements of the protocol
* A subject previously enrolled in study NCT00294047, who received the control vaccine, and who cannot receive the GSK580299 vaccine because the subject is above the age for which the vaccine is licensed.
* Written informed consent obtained from the subject
* Free of obvious health problems as established by medical history and clinical examination before entering into the study.
* Female subjects of non-childbearing potential may be enrolled in the study.
* Female subjects of childbearing potential may be enrolled in the study, if the subject:

  * has practiced adequate contraception for 30 days prior to vaccination, and
  * has a negative pregnancy test on the day of vaccination, and
  * has agreed to continue adequate contraception during the entire treatment period and for 2 months after completion of the vaccination series.

Exclusion Criteria:

* Pregnant or breastfeeding.
* A women planning to become pregnant, likely to become pregnant or planning to discontinue contraceptive precautions during the vaccination phase of the study, i.e. up to two months after the last vaccine dose.
* Use of any investigational or non-registered product other than the study vaccine within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Previous vaccination against HPV or planned administration of another HPV vaccine during the study other than that foreseen in the protocol.
* Chronic administration of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose. For corticosteroids, this will mean prednisone greater than or equal to 20 mg/day, or equivalent. Inhaled and topical steroids are allowed
* Planned administration/administration of a vaccine not foreseen by the study protocol within 30 days (i.e., Day 0-29) of each dose of vaccine, with the exception of administration of routine meningococcal, hepatitis B, hepatitis A, inactivated influenza, diphtheria/tetanus and/or diphtheria/tetanus-containing vaccine up to 8 days before each dose of study vaccine. Enrolment will be deferred until the subject is outside of specified window.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product.

NOTE: Subjects enrolled in this study may also be eligible for a four-year gynaecological follow-up of the HPV-015 study, in which no investigational product will be administered. Subjects will be invited to the gynaecological follow-up study if either of the following applies:

* if they test positive for oncogenic HPV infection, but display normal cervical cytology at their concluding HPV-015 study end visit;
* if they are pregnant so that no cervical sample can be taken at their concluding HPV-015 study end visit;

  * Previous administration of any components of the vaccine.
  * Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
  * Cancer or autoimmune disease under treatment.
  * Administration of immunoglobulins and/or any blood products within the 3 months preceding the first dose of study vaccine or planned administration during the study period.
  * History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccine
  * History of any neurological disorders or seizures.
  * Acute disease and/or fever at the time of enrolment.
  * Acute or chronic, clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by physical examination or laboratory screening tests.

Min Age: 26 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2011-04-01 (Actual); Primary Completion 2017-11-23 (Actual); Study Completion 2017-11-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (26):
- United States (19):
  - GSK Investigational Site, Aurora, Colorado
  - GSK Investigational Site, Golden, Colorado
  - GSK Investigational Site, Coral Gables, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Augusta, Georgia
  - GSK Investigational Site, Iowa City, Iowa
  - GSK Investigational Site, Wichita, Kansas
  - GSK Investigational Site, Bardstown, Kentucky
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Lebanon, New Hampshire
  - GSK Investigational Site, New Bern, North Carolina
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Carnegie, Pennsylvania
  - GSK Investigational Site, Erie, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Salt Lake City, Utah
  - GSK Investigational Site, Wenatchee, Washington
- Canada (7):
  - GSK Investigational Site, Edmonton, Alberta
  - GSK Investigational Site, Vancouver, British Columbia
  - GSK Investigational Site, Halifax, Nova Scotia
  - GSK Investigational Site, Truro, Nova Scotia
  - GSK Investigational Site, Waterloo, Ontario
  - GSK Investigational Site, Québec, Quebec
  - GSK Investigational Site, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: Yes
IPD is available via the Clinical Study Data Request site (click on the link provided below)
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months
URL: http://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted by multiple investigators at 28 centers in Canada and the United States.
Pre-assignment Details: All subjects enrolled were vaccinated and included in the Total Vaccinated cohort (TVc).
Period: Overall Study
Arm/Group | Cervarix Group
Started | 137
Completed | 131
Not Completed | 6
Not completed — Lost to Follow-up | 4
Not completed — Withdrawal by Subject | 1
Not completed — Migrated/moved from study area | 1

BASELINE CHARACTERISTICS:
Arm/Group | Cervarix Group
Number analyzed (Participants) | 137
Age, Continuous [Mean (Standard Deviation); unit: Years] | 47.9 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 137
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Geographic Ancestry: African Heritage/African American | 11
  Geographic Ancestry: Asian - East Asian Heritage | 1
  Geographic Ancestry: Asian - Japanese Heritage | 2
  Geographic Ancestry: White - Arabic/North African Heritage | 1
  Geographic Ancestry: White - Caucasian/European Heritage | 119
  Geographic Ancestry: Native Canadian | 2
  Geographic Ancestry: Cuban | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Serious Adverse Events (SAEs)
Description: Assessed SAEs included medical occurrences that resulted in death, were life-threatening, required hospitalization or prolongation of hospitalization, resulted in disability/incapacity or were congenital anomalies/birth defects in the offspring of a study subject. Any SAE = occurrence of the SAE regardless of intensity grade. Grade 3 SAE = an SAE which prevented normal, everyday activities. Related SAE = an SAE assessed by the investigator as causally related to the study vaccination.
Time Frame: During the entire study period (from Day 0 up to Month 12)
Population: The analysis was performed on the Total Vaccinated cohort (TVc), which included all vaccinated subjects for whom safety data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group
Number analyzed (Participants) | 137
Participants
  Any SAE(s) | 1
  Grade 3 SAE(s) | 1
  Related SAE(s) | 0

2. Primary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Medically Significant Conditions (MSCs)
Description: Medically significant conditions were defined as: AEs prompting emergency room or physician visits that were not (1) related to common diseases, or (2) not related to routine visits for physical examination or vaccination, or as SAEs that were not related to common diseases. Common diseases included: upper respiratory infections, sinusitis, pharyngitis, gastroenteritis, urinary tract infections, cervicovaginal yeast infections, menstrual cycle abnormalities and injury. Any MSC = occurrence of the MSC regardless of intensity grade. Grade 3 MSC = a MSC which prevented normal, everyday activities. Related MSC = MSC assessed by the investigator as related to the study vaccination.
Time Frame: During the entire study period (from Day 0 up to Month 12)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group
Number analyzed (Participants) | 137
Participants
  Any MSC(s) | 24
  Grade 3 MSC(s) | 2
  Related MSC(s) | 1

3. Primary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Potentially Immune-Mediated Diseases (pIMDs)
Description: pIMD(s) are a subset of medically significant conditions (MSCs) that included autoimmune diseases and other inflammatory and/or neurological disorders of interest which may or may not have had an autoimmune aetiology. Any pIMD = occurrence of the pIMD regardless of intensity grade. Grade 3 pIMD = a pIMD which prevented normal, everyday activities. Related pIMD = pIMD assessed by the investigator as related to the study vaccination.
Time Frame: During the entire study period (from Day 0 up to Month 12)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group
Number analyzed (Participants) | 137
Participants
  Any pIMD(s) | 1
  Grade 3 pIMD(s) | 0
  Related pIMD(s) | 0

4. Primary Outcome: Number of Subjects Reporting Pregnancies and Outcomes of the Reported Pregnancies
Description: Pregnancy is the term used to describe the period in which a fetus develops inside a woman's womb or uterus. In this study, the number of subjects with pregnancies was calculated. The subjects with confirmed pregnancies were followed up to determine the outcomes of the reported pregnancies.
Time Frame: During the entire study period (from Day 0 up to Month 12)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group
Number analyzed (Participants) | 137
Participants | 0

ADVERSE EVENTS:
Time Frame: During the entire study period (from Day 0 up to Month 12).
Arm/Group | Cervarix Group
All-Cause Mortality (participants affected / at risk) | 0/137
Serious Adverse Events (participants affected / at risk) | 1/137
Other Adverse Events (participants affected / at risk) | 24/137
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cervarix Group (N=137)
Menorrhagia (Reproductive system and breast disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cervarix Group (N=137)
Anaemia (Blood and lymphatic system disorders) | 2 (2)
Anxiety (Psychiatric disorders) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Chloasma (Skin and subcutaneous tissue disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
Complex regional pain syndrome (Nervous system disorders) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 1 (1)
Conjunctivitis allergic (Eye disorders) | 1 (1)
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Crohn's disease (Gastrointestinal disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Furuncle (Infections and infestations) | 1 (1)
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 1 (1)
Mastitis (Infections and infestations) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Otitis media (Infections and infestations) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 2 (2)
Pneumonia (Infections and infestations) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 1 (1)
Skin burning sensation (Skin and subcutaneous tissue disorders) | 1 (1)
Staphylococcal infection (Infections and infestations) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1)
Ulnar nerve injury (Injury, poisoning and procedural complications) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2011-01-13): https://cdn.clinicaltrials.gov/large-docs/89/NCT01190189/Prot_000.pdf
  • Statistical Analysis Plan (2015-09-25): https://cdn.clinicaltrials.gov/large-docs/89/NCT01190189/SAP_001.pdf